CLINICAL TRIAL: NCT02985372
Title: Efficacy and Safety of Decitabine in Combination With Low-dose Cytarabine as Inductive Treatment in Newly Diagnosed Elderly Patients With Acute Myeloid Leukemia
Brief Title: Decitabine in Combination With Low-dose Cytarabine in Elderly Patients With Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chunyan Ji (Other)
Collaborators: Binzhou Medical University (Other); Shengli Oilfield Hospital (Other); Heze Municipal Hospital (Other); Jinan Military Genaral Hospital (Unknown); Jinan Central Hospital (Other); Jining Medical University (Other); Linyi People's Hospital (Other); Qingdao University (Other); Rizhao People's Hospital (Other); Qianfoshan Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other); Taian City Central Hospital (Other); Taishan Medical University Affiliated Hospital (Other); Weihai Municipal Hospital (Other); Weifang Medical University (Other); Zibo First Hospital (Other); Central Hospital of Zibo (Other)
Responsible Party: Sponsor-Investigator, Chunyan Ji, professor, Shandong University
Organization: Shandong University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESDCLDC in NDEAML
Record Dates: First submitted 2016-11-25; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-11

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute myeloid leukemia (Experimental): All patients were treated with decitabine of 15 mg/ m2 intravenously over 4h for 5 consecutive days (day 1-5) for priming combined with cytarabine of 10 mg/m2 q12h for 10 days (day 4-13).
  Interventions: Drug: Decitabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Decitabine — All patients were treated with decitabine of 15 mg/ m2 intravenously over 4h for 5 consecutive days (day 1-5) for priming combined with cytarabine of 10 mg/m2 q12h for 10 days (day 4-13).
Drug: Cytarabine

SUMMARY:
This prospective multicenter clinical study was designed to assess the efficacy and safety of decitabine in combination with low-dose cytarabine induction treatment for elderly patients with newly diagnosed acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
All patients were treated with decitabine of 15 mg/ m2 intravenously over 4h for 5 consecutive days (day 1-5) for priming combined with cytarabine of 10 mg/m2 q12h for 10 days (day 4-13).

Hydroxyurea was permitted as rescue medication if white blood count (WBC) was >20×109/L and but was discontinued at least 24h before decitabine treatment.

Supportive care including blood product transfusions, G-CSF, antiemetic medications, antiviral and antifungal medications, or empiric antibiotics may be used at the clinical discretion of the investigator.

Curative effect was evaluated after two cycles:

1. <5% blast in the marrow, enter into maintenance therapy (Group A)
2. ≥5% blast in the marrow, continue induction therapy two cycles,

   ① <5% blast in the marrow, enter into maintenance therapy (Group B);

   ② ≥5% blast in the marrow, dropped out of the study (Group C)
3. marrow blast decline <60%, dropped out of the study (Group C).

Maintenance therapy regimen:

1. Ara-C 1g/m2/d iv drip d1-4 1 cycle
2. DEC 15mg/m2/d iv drip d1-5 1 cycle
3. Ara-C 1g/m2/d iv drip d1-4 1 cycle
4. DEC 15mg/m2/d iv drip d1-5 1 cycle

ELIGIBILITY:
Inclusion Criteria:

1. Patients with previously untreated non-M3 AML (diagnosed by the WHO2016 criteria).
2. Age: ≥ 60 and ≤ 75 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5x upper limit of normal (ULN), total bilirubin ≤ 1.5 ULN, serum creatinine < 2ULN.
5. Without central nervous system symptoms.
6. Willing to accept the follow-up.
7. Normal heart function(EF>50%). The subjects volunteer to sign the informed consent.

Exclusion Criteria:

1. With severe cardiac, renal or hepatic insufficiency.
2. With other cancers requiring treatment.
3. With other hematological diseases(e.g. Hemophilia, myelofibrosis, etc.).
4. With severe infection or metabolic disease(including tuberculosis and pulmonary aspergillosis).
5. Brain disorders or severe mental diseases which could limit compliance with study requirements.
6. Major operation within 3 weeks.
7. With HIV infection or AIDS-associated diseases.
8. Any drug abuse, medical, mental or social situations which would affect the results.
9. Hypersensitivity to cytarabine (not including drug fever or exanthema) or decitabine.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | three years
complete remission rate | three years

SECONDARY OUTCOMES:
Overall survival | three years
progression-free survival | three years
mortality rate | three years
recurrence rate | three years

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ji, Doctor, Study Chair — Shandong University

IPD SHARING:
Plan to Share IPD: Undecided